CLINICAL TRIAL: NCT07404943
Title: The Effect of Telenursing Counseling on Functioning and Treatment Adherence Levels in Individuals With Bipolar Disorder
Brief Title: The Effect of Telenursing on Functionality and Treatment Adherence in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Ayhan (Other)
Responsible Party: Sponsor-Investigator, Didem Ayhan, Assoc. prof, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-257
Record Dates: First submitted 2026-01-24; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Bi-Polar Disorder
Keywords: bi-polar; Treatment Adherence; Functioning; telenursing
MeSH Terms: conditions — Bipolar Disorder; Treatment Adherence and Compliance | interventions — Telenursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): group receiving telenursing counseling
  Interventions: Behavioral: telenursing
- control group (No Intervention): group receiving routine community mental health care

INTERVENTIONS:
Behavioral: telenursing — Providing nursing services by telephone is not standard practice in community mental health centers.
  Arms: experimental group

SUMMARY:
This research is a randomized controlled experimental study with a pretest-posttest design, conducted to determine the effect of telenursing counseling on functionality and treatment adherence levels in patients with bipolar disorder.

First, patients followed up with a diagnosis of bipolar disorder at the Community Mental Health Center (CMHC) were evaluated by the researcher through face-to-face interviews in terms of the inclusion criteria. Patients who met the criteria and voluntarily agreed to participate in the study were informed about the research, and their written informed consent was obtained. Subsequently, the participants were assigned to the experimental and control groups by an independent faculty member using a stratified block randomization method. Following the randomization process, a nurse working at the Community Mental Health Center administered the Descriptive Information Form, the Short Functioning Assessment Scale, and the Morisky Medication Adherence Scale to both groups face-to-face as a pretest.

After the baseline measurements, an eight-week telenursing counseling intervention was implemented with the patients in the experimental group. No intervention was provided to the control group; they only received standard treatment and care services. At the end of the eight-week period, the same nurse working at the CMHC administered the SFAS and MMAS scales again, and the posttest measurements were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Having received a diagnosis of bipolar disorder (Type I/II) at least one year ago according to the diagnostic criteria specified in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR),
* Being followed up at the Community Mental Health Center (CMHC) for at least one year,
* Having a Morisky Medication Adherence Scale score of ≥ 1,
* Having at least a primary school education,
* Owning a mobile phone and having no visual and/or hearing impairment related to calling/messaging use,
* Voluntarily agreeing to participate in the research.

Exclusion Criteria:

* Presence of an acute mood episode,
* Presence of a comorbid mental disorder (e.g., severe personality disorder, substance use disorder),
* Being unable to continue tele-intervention due to a serious physical illness (e.g., cancer, heart failure) and/or cognitive impairment (e.g., loss of intellectual capacity, neurocognitive disorder),
* Presence of conditions that make tele-access impossible,
* Concurrent participation in another psychoeducation or tele-intervention program with similar content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of experimental and control groups and comparison of pre-test and post-test results for Morisky Medication Adherence Scale | From the registration phase to the end of the 8-week telenursing program
  Morisky Medication Adherence Scale: The scale items are answered as "yes (1 point)" and "no (0 points)". The total score obtainable from the scale ranges from 0 to 4. Accordingly, a score of 0 indicates high medication adherence, 1-2 points indicate medium adherence, and 3-4 points indicate low adherence.
Comparison of experimental and control groups and comparison of pre-test and post-test results for Short Functioning Assessment Scale | From the registration phase to the end of the 8-week telenursing program
  Short Functioning Assessment Scale (SFAS): The scale consists of 24 items on a four-point Likert scale ("0: no difficulty", "1: minimal difficulty", "2: moderate difficulty", "3: severe difficulty"). SFAS has six subscales: autonomy, occupational functioning, cognitive functioning, financial matters, interpersonal relationships, and leisure activities. The total score on the scale ranges from 0 to 72, with higher scores indicating poorer functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Evliya Çelebi Training and Research Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual assessments will not be conducted; analyses will be based on the total number.

REFERENCES:
- [Background] Raesi R, Shaye ZA, Saghari S, Sheikh Beig Goharrizi MA, Raei M, Hushmandi K. The impact of education through nurse-led telephone follow-up (telenursing) on the quality of life of COVID-19 patients. J Egypt Public Health Assoc. 2021 Nov 8;96(1):30. doi: 10.1186/s42506-021-00093-y. PMID 34748085
- [Background] Oz HS, Ayhan D, Oz F. Effects of Telenursing on Drug Attitudes, Self-Efficacy, and Quality of Life in Individuals With Schizophrenia: A Randomized Controlled Trial. J Psychosoc Nurs Ment Health Serv. 2024 Oct;62(10):15-24. doi: 10.3928/02793695-20240423-02. Epub 2024 May 6. PMID 38709104
- [Background] Van der Walt JP, Scott DB. Bullera dendrophila sp. n. Antonie Van Leeuwenhoek. 1970;36(3):383-7. doi: 10.1007/BF02069038. No abstract available. PMID 5312514
- [Background] Nierenberg AA, Agustini B, Kohler-Forsberg O, Cusin C, Katz D, Sylvia LG, Peters A, Berk M. Diagnosis and Treatment of Bipolar Disorder: A Review. JAMA. 2023 Oct 10;330(14):1370-1380. doi: 10.1001/jama.2023.18588. PMID 37815563
- [Background] Najafi SS, Shaabani M, Momennassab M, Aghasadeghi K. The Nurse-Led Telephone Follow-Up on Medication and Dietary Adherence among Patients after Myocardial Infarction: A Randomized Controlled Clinical Trial. Int J Community Based Nurs Midwifery. 2016 Jul;4(3):199-208. PMID 27382586
- [Background] Miller JN, Black DW. Bipolar Disorder and Suicide: a Review. Curr Psychiatry Rep. 2020 Jan 18;22(2):6. doi: 10.1007/s11920-020-1130-0. PMID 31955273
- [Background] Miklowitz DJ, Efthimiou O, Furukawa TA, Scott J, McLaren R, Geddes JR, Cipriani A. Adjunctive Psychotherapy for Bipolar Disorder: A Systematic Review and Component Network Meta-analysis. JAMA Psychiatry. 2021 Feb 1;78(2):141-150. doi: 10.1001/jamapsychiatry.2020.2993. PMID 33052390